CLINICAL TRIAL: NCT06608433
Title: Glucagon-like Peptide-1 Receptor Agnoists for the Assessment of Adrenal Function - the PIANO Study
Brief Title: Glucagon-like Peptide-1 Receptor Agnoists for the Assessment of Adrenal Function
Acronym: PIANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: EKNZ2024-01744
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteer Study; HPA; Cortisol Deficiency; Adrenal Insufficiency
Keywords: Hypothalamo-pituitary-adrenal axis; Healthy volunteers; Glucagon-like peptide-1 receptor agonists; GLP-1 receptor agnoists; semaglutide; adrenal insufficiency; HPA axis; adrenal function testing
MeSH Terms: conditions — Adrenal Insufficiency | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide/Rybelsus (Experimental)
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: semaglutide — semaglutide/Rybelsus will be administered as a single oral dose
  Arms: Semaglutide/Rybelsus
Drug: Placebo — Placebo pills will be administered as a single oral dose
  Arms: Placebo

SUMMARY:
This study aims to investigate the effects of a single dose of the glucagon-like 1 receptor agonist semaglutdie/Rybelsus on the hypothalamo-pituitary-adrenal axis, thus cortisol levels and other stresshormones in healthy males.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18-60 years
* BMI 18.5-30 kg/m2
* No regular medication

Exclusion Criteria:

* participation in a trial with investigational drugs within 30 days
* vigorous physical exercise within 24 hours before the study participation
* alcohol intake within 24 hours before the study participation
* a history of intake of glucocorticoids or GLP-1 RA within the last 8 weeks.
* Known allergy towards GLP-1 RA

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in serum cortisol after Rybelsus vs. Placebo | within 210 minutes after the intake of the study drug
  The primary endpoint is the difference between the two visits (placebo vs. Rybelsus) in the change in cortisol from cortisol baseline to the maximally stimulated cortisol value (cortisolmax).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No